CLINICAL TRIAL: NCT04809259
Title: Ambulatory Administration of Meropenem With Elastomeric Pumps and an Isothermal Pouch
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Serge de Valliere, Physician, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Meropenem 2021
Record Dates: First submitted 2021-02-03; First posted 2021-03-22 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Infection, Bacterial
Keywords: Meropenem; Outpatient parenteral antimicrobial therapy; Elastomeric pumps; Continuous infusion
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous infusion of meropenem (Experimental): The meropenem solution will be administered continuously using elastomeric pumps which will be changed every 24 hours and which will be inserted in an isothermal pouch to ensure that the antibiotic solution is maintained at a temperature between 10° and 15°
  Interventions: Device: Isothermal pouch

INTERVENTIONS:
Device: Isothermal pouch — The study will verify it the use of an isothermal pouch to maintain the content of an elastomeric pump at 10° to 15°C avoids unacceptable meropenem degradation over the 24 hour infusion period.

SUMMARY:
This study aims to evaluate if meropenem can be administered in outpatients as a continuous infusion using elastomeric pumps and an isothermal pouch maintaining the anti-infective solution between 10° and 15°C for improved stability.

DETAILED DESCRIPTION:
The Outpatient Parenteral Antibiotic Therapy (OPAT) unit of the University Hospital of Lausanne uses elastomeric pumps for continuous intravenous administration of 6 different antibiotics. This mode of administration is possible for all antibiotics with a time-dependent bactericidal effect.

Meropenem belongs to this class of antibiotics, but is not stable at room temperature in elastomeric pumps. However, this antibiotic is stable at 10°C and 15°C. The investigators have therefore developed an isothermal pouch that allows the anti-infective solution to be maintained at a temperature between 10 and 15°C over 24 hours.

This study aims to evaluate the efficacy and safety of meropenem administration using an elastomeric pump maintained at a temperature between 10° and 15°C by an isothermal pouch.

The possibility of being able to administer meropenem by elastomeric pumps would greatly facilitate the ambulatory management of patients requiring treatment with this anti-infective drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the OPAT unit for a anti-microbial treatment with meropenem
* Age ≥ 18 years
* Informed consent signed

Exclusion Criteria:

* Patients refusing a PICC-line
* Pregnancy or desire of a pregnancy
* Patients considered to be not eligible for outpatient treatment by the OPAT team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of plasma meropenem levels ≥ 4 mg/L | Will be determined at 24 hours, and then every 72 to 96 hours through treatment completion
  Blood will be drawn to determine meropenem plasma concentrations

SECONDARY OUTCOMES:
Cure or stabilisation of infection | 3 months after beginning of treatment
  Number of patients who are cured or have a stabilisation of the infection
Readmission | 3 months after beginning of treatment
  Number of patients who are unexpectedly readmitted to hospital
Allergic reactions or abnormal blood tests | Once a week through treatment completion
  Number of patients who develop an allergic reaction or abnormal blood results, which will include full blood count, creatinine, alanine-aminotransferase (ALT)
Volume administered by elastomeric pumps | Will be determined at 24 hours, and then every 72 to 96 hours through treatment completion
  Residual fluid volume in the elastomeric pumps
Meropenem concentration in elastomeric pumps | Will be determined at 24 hours, and then every 72 to 96 hours through treatment completion
  Measurement of meropenem concentration in the elastomeric pumps

CONTACTS AND LOCATIONS:
Overall Officials: Serge de Vallière, Principal Investigator — de Vallière Serge

IPD SHARING:
Plan to Share IPD: No